CLINICAL TRIAL: NCT01685775
Title: Needlescopic Versus Transvaginal/Transumbilical Cholecystectomy: a Randomized Clinical Trial
Brief Title: Needlescopic Versus Transvaginal/Transumbilical Cholecystectomy
Acronym: NATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Dirk R. Bulian, Principal Investigator, University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1114-7386; DRKS00000341 (Registry Identifier: DRKS-ID)
Record Dates: First submitted 2012-09-04; First posted 2012-09-14 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Calculus of Gallbladder With or Without Cholecystitis; Laparoscopic Cholecystectomy
Keywords: Gallbladder; cholecystectomy; NOTES; natural orifice transluminal endoscopic surgery; gallstone
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transvaginal/transumbilical cholecystectomy (Experimental): Transvaginal/transumbilical group: we will use a 5 mm trocar in the umbilicus and a 10 mm trocar together with a 5 mm seizing forceps through the posterior vaginal vault to perform the cholecystectomy in the Zornig style
  Interventions: Procedure: Transvaginal/transumbilical
- Needlescopic cholecystectomy (Active Comparator): Needlescopic cholecystectomy with 3 trocars: we will use two 2-3 mm working trocars and one 10 mm optic trocar, its access is also used for extraction of the gallbladder
  Interventions: Procedure: Needlescopic with 3 trocars

INTERVENTIONS:
Procedure: Transvaginal/transumbilical
  Arms: Transvaginal/transumbilical cholecystectomy
Procedure: Needlescopic with 3 trocars
  Arms: Needlescopic cholecystectomy

SUMMARY:
Laparoscopic surgery has become the golden standard for the removal of the gallbladder. Recently, developments have been made so that operations can be performed through a natural orifice instead of the abdominal wall, thus minimizing the trauma of a procedure. This study compares the transvaginal/transumbilical cholecystectomy with the laparoscopic operation using 2-3mm instruments in female patients. It also examines the benefits and disadvantages related to postoperative pain, cosmetic aspects, and potential physiological alterations to the transvaginal approach that affect sexual intercourse.

DETAILED DESCRIPTION:
The amount of trauma inflicted, especially in abdominal operations, depends largely on target organ access. Great efforts have been made to minimize access trauma. The further development of laparoscopy led to the miniaturization of surgical instruments and otherwise the use of natural orifices, like the stomach, rectum or vagina. The cholecystectomy is currently performed needlescopicly with 2-3 mm trocars and in transumbilically assisted transvaginal technique. The aim of this randomized study is to compare these two techniques in female patients that are in need of an elective cholecystectomy. The patients will be randomized on a 1:1 ratio into two treatment groups. In the needlescopic group the investigators will use two 2-3 mm working trocars and one 10 mm optic trocar, also to extract the gallbladder. In the transvaginal/transumbilical group the investigators will perform the Zornig technique using a 5 mm trocar in the umbilicus and a 10 mm trocar together with a 5 mm seizing forceps through the posterior vaginal vault. The primary endpoint of this trial is to measure the intensity of pain in motion measured from the day of the operation until postoperative day 2. Four different measurements of pain will be used. Furthermore the investigators examine perioperative complications as security parameters. The trial is supported in part by the German Ministry of Research and Education (CHIR-Net grant, BMBF No. 01-GH-0605).

ELIGIBILITY:
Inclusion Criteria:

* Gender: Female
* Minimum Age: 18 Years
* Maximum Age: 80 Years
* indication for elective cholecystectomy on account of symptomatic cholecystolithiasis
* age >=18 years and <=80 years
* legal competence

Exclusion Criteria:

* Acute cholecystitis or locally complicated disease (gallbladder empyema, choledocholithiasis, pancreatitis, etc.)
* liver cirrhosis (Child Pugh A, B, C)
* severe comorbidity, class IV or V as defined by the American Society for Anesthesiologists (ASA)
* intact hymen
* acute vaginal infection
* lacking visibility of the uterine orifice
* endometriosis
* malignoma
* obesity with a Body Mass Index (BMI) > 40 kg/m2
* chronic abuse of analgesics or alcohol
* neuromuscular disease that could interfere treatment or measures of pain
* history of major abdominal surgery with a high risk of intraperitoneal adhesions (minor operations such as an appendectomy, inguinal hernia repair, minor gynaecological surgery, etc. will not be considered exclusion criteria)
* gravidity or breastfeeding
* allergy against analgesics
* patients who are dependent on or employed by the trial sponsor or physicians
* institutionalisation for legal reasons
* participation in other clinical studies that could interfere with the present trial
* no written informed consent signed

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Intensity of pain in motion | at the operation day
  Pain Scores on the Visual Analog Scale (0-10)
Intensity of pain in motion | at postoperative day 1
  2 measures (in the morning and in the evening) Pain Scores on the Visual Analog Scale (0-10)
Intensity of pain in motion | at postoperative day 2
  Pain Scores on the Visual Analog Scale (0-10)

SECONDARY OUTCOMES:
Cosmetic aspects and overall satisfaction with the results of the surgery | 10 days after operation
  1 (complete satisfaction) to 5 (complete dissatisfaction) scale from patient's and surgeon's point of view
Intraoperative complications | evaluated at the operation day
  e.g. bleeding, organ-injury, especially bile-duct-injury
Duration of the operation | at the operation day
  (in minutes)
Surgical handling for the first and second surgeon | evaluated at the operation day
  on a 1 to 5 scale
Intensity of pain in motion | at postoperative day 2
  in the evening pain Scores on the Visual Analog Scale (0-10)
Cumulative use of analgesics | 10 days after the surgery
  quantity, dose and class of the used drugs
Return to everyday, work related and free time activities | 3 months after operation
  duration of limitations.
Quality of life | on postoperative day 10
  measured with the Gastrointestinal Quality of Life Index (GIQLI) from Eypasch et al.
Postoperative restrictions of sexual function | 3 months after surgery
  with questions 14-19 of the "female sexual function index" (FSFI-D)
Morphological consequences of transvaginal access | at the day before the operation, and again 10 to 14 days and 6 months after their surgery
  all patients from the transvaginal/transumbilical group will be examined by a gynaecologist
Cosmetic aspects and overall satisfaction with the results of the surgery | 3 months after operation
  1 (complete satisfaction) to 5 (complete dissatisfaction) scale from patient's and surgeon's point of view
Cosmetic aspects and overall satisfaction with the results of the surgery | 6 months after operation
  1 (complete satisfaction) to 5 (complete dissatisfaction) scale; from patient's and surgeon's point of view
Conversionrate | at the operation day
  Conversion from transvaginal to classical laparoscopic or open technique and from needlescopic to open technique
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | at 6 month
  including frequency of reoperation
Intensity of pain in motion | at postoperative day 3
  in the morning and in the evening pain Scores on the Visual Analog Scale (0-10)
Intensity of pain in motion | at postoperative day 4
  in the morning and in the evening pain Scores on the Visual Analog Scale (0-10)
Intensity of pain in motion | at postoperative day 5
  in the morning and in the evening pain Scores on the Visual Analog Scale (0-10)
Intensity of pain in motion | at postoperative day 6
  in the morning and in the evening pain Scores on the Visual Analog Scale (0-10)
Intensity of pain in motion | at postoperative day 7
  in the morning and in the evening pain Scores on the Visual Analog Scale (0-10)
Intensity of pain in motion | at postoperative day 8
  in the morning and in the evening pain Scores on the Visual Analog Scale (0-10)
Intensity of pain in motion | at postoperative day 9
  in the morning and in the evening pain Scores on the Visual Analog Scale (0-10)
Intensity of pain in motion | at postoperative day 10
  in the morning and in the evening pain Scores on the Visual Analog Scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk R. Bulian, Principal Investigator — Witten/Herdecke University
Locations (1):
- Department of Abdominal, Vascular and Transplant Surgery; Cologne-Merheim Medical Center, Cologne, Germany

REFERENCES:
- [Background] Bulian DR, Trump L, Knuth J, Siegel R, Sauerwald A, Strohlein MA, Heiss MM. Less pain after transvaginal/transumbilical cholecystectomy than after the classical laparoscopic technique: short-term results of a matched-cohort study. Surg Endosc. 2013 Feb;27(2):580-6. doi: 10.1007/s00464-012-2490-2. Epub 2012 Aug 28. PMID 22926893
- [Background] Bulian DR, Trump L, Knuth J, Cerasani N, Heiss MM. Long-term results of transvaginal/transumbilical versus classical laparoscopic cholecystectomy--an analysis of 88 patients. Langenbecks Arch Surg. 2013 Apr;398(4):571-9. doi: 10.1007/s00423-013-1071-8. Epub 2013 Mar 1. PMID 23456357
- [Result] Bulian DR, Knuth J, Cerasani N, Sauerwald A, Lefering R, Heiss MM. Transvaginal/transumbilical hybrid--NOTES--versus 3-trocar needlescopic cholecystectomy: short-term results of a randomized clinical trial. Ann Surg. 2015 Mar;261(3):451-8. doi: 10.1097/SLA.0000000000000218. PMID 24108196